CLINICAL TRIAL: NCT00847756
Title: Thorough Clinical Investigation of the Host-pathogen Interaction in Chronic and Recurrent Otitis Media
Brief Title: Host-pathogen Interaction in Otitis Media
Acronym: OMVac
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Prof. dr. R. de Groot, head department of Pediatrics, Radboud University Nijmegen Medical Centre, Nijmegen, the Netherlands
Other Study IDs: OMVac clinical study; EU-FP6 (Registry Identifier: 037653)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2010-12

CONDITIONS: Otitis Media
Keywords: Otitis media; demography; Streptococcus pneumoniae; Haemophilus influenzae; Moraxella catarrhalis; rhinovirus; children, 0-5 years of age; diagnosed rAOM, COME or CSOM by an otorhinolaryngologist; primary and secondary hospital Nijmegen, the Netherlands
MeSH Terms: conditions — Otitis Media; Haemophilus Infections | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood nasopharyngeal swab middle ear fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- rAOM: Children 0-5 years of age suffering from recurrent acute otitis media and waiting for tympanostomy tube insertion.
  Interventions: Other: questionnaire; Procedure: blood sample; Procedure: collection of middle ear fluid; Procedure: nasopharyngeal swab
- COME: Children 0-5 years of age suffering from chronic otitis media with effusion and waiting for tympanostomy tube insertion.
  Interventions: Other: questionnaire; Procedure: blood sample; Procedure: collection of middle ear fluid; Procedure: nasopharyngeal swab
- CSOM: Children 0-5 years of age suffering from chronic suppurative otitis media and waiting for tympanostomy tube insertion. Note: Only 3 patients with CSOM were recruited and therefore not suitable for publication.

INTERVENTIONS:
Other: questionnaire — Identification of risk factors
  Groups: COME; rAOM
Procedure: blood sample — venal puncture, 5ml. A blood sample will be taken at the day of surgery and after 2-3 months.
  Groups: COME; rAOM
Procedure: collection of middle ear fluid — During routine surgery middle ear fluids are collected per patient.
  Groups: COME; rAOM
Procedure: nasopharyngeal swab — A nasopharyngeal swab is taken at the end of the surgical procedure and after 2-3 months.
  Groups: COME; rAOM

SUMMARY:
Otitis Media (OM) is one of the most frequent diseases in childhood and the primary reason for children to visit a physician. In many countries it is the most common reason to prescribe antibiotics leading to increased drug-resistance of the causative agents, or to undergo surgery. Costs for general health care are expanding, and are estimated to be 3-5 billion dollar annually in the United States. Prevention is suspected to be an important solution to this problem.

Although OM management has no universal standard yet, it may imply watchful waiting, antibiotic treatment, adenoidectomy, insertion of tympanostomy tubes and (future) vaccination. Approximately 80% of the acute otitis media (AOM) cases is self-limiting within 2-14 days and also otitis media with effusion (OME) resolves spontaneously: 60% of newly detected OME resolves within 3 months. However, in a significant part of the OM population persistent or recurrent episodes of OM are responsible for a significant morbidity for both children and parents, despite variable treatment options.

Through the set up of a new prospective cohort in a clinical setting, relevant patient characteristics, the role of bacterial and viral pathogens, the role of recurrent infection in relation to biofilm formation, and the host response at protein level will be studied in detail. This project is expected to increase the understanding of the underlying mechanisms of OM disease, which will support future treatment and prevention strategies. Better understanding in OM pathogenesis is warranted in order to develop these novel preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* children up to 5 years of age
* suffering from rAOM, COME or CSOM
* waiting for tympanostomy tube insertion
* informed consent

Exclusion Criteria:

* No informed consent
* The child has a malignancy, or organ transplantation, or immune deficiency in the medical history
* The child had recent elective ear surgery (i.e. mastoidectomy, implants <2 weeks ago)
* The child suffers from systemic infectious diseases (i.e. hepatitis, chickenpox)

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children up to 5 years of age suffering from rAOM, COME or CSOM waiting for tympanostomy tube insertion
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Detection of biological markers in blood which inform us about the risk of recurrent infection and severity of disease | 01-06-2009 to 01-06-2010

SECONDARY OUTCOMES:
Otitis media demography | 15-04-2008 to 01-01-2010
Bacterial and viral pathogen detection | 15-04-2008 to 01-01-2010
Determination of the molecular and cellular immune response in relation to viral and bacterial pathogens | 15-04-08 to 01-01-2010
Gene expression profiling of the three major bacterial pathogens: S. pneumoniae, H. influenzae and M. catarrhalis | 01-06-2009 to 01-06-2010

CONTACTS AND LOCATIONS:
Overall Officials: Ronald de Groot, MD, PhD, Study Chair — Department of Pediatrics, Radboud University Nijmegen Medical Centre, Nijmegen, the Netherlands; Kim Stol, MD, Principal Investigator — Department of Pediatrics, Radboud University Nijmegen Medical Centre, Nijmegen, the Netherlands
Locations (2):
- Netherlands (2):
  - Canisius Wilhelmina hospital, Department of otorhinolaryngology, Nijmegen
  - Radboud, University Nijmegen Medical Centre, Department of Otorhinolaryngology, Nijmegen